CLINICAL TRIAL: NCT00771771
Title: Early Supported Discharge After Stroke in Bergen. An RCT Looking at the Collaboration Between Hospital Service and Primary Health Care.
Brief Title: Early Supported Discharge After Stroke in Bergen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: University of Bergen (Other); Municipality of Bergen, Norway (Unknown); Kavli Research Centre for Ageing and Dementia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18993
Record Dates: First submitted 2008-10-10; First posted 2008-10-13 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Stroke
Keywords: Stroke; Rehabilitation; Early Supported Discharge; ESD; RCT
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Day unit rehabilitation (Active Comparator): Discharge from the hospital to the patients' homes as soon as possible, supported by an out-patient ambulatory coordinating multidisciplinary team. The patients will be offered rehabilitation in a day unit, and multidisciplinary policlinical follow-ups will be performed 3 and 6 months after inclusion.
  Interventions: Other: Early supported discharge with day unit rehabilitation
- Home rehabilitation (Active Comparator): Discharge from the hospital to the patients' homes as soon as possible, supported by an out-patient ambulatory coordinating multidisciplinary team. The patients will be offered rehabilitation treatment in their homes, and multidisciplinary policlinical follow-ups will be performed 3 and 6 months after inclusion.
  Interventions: Other: Early supported discharge with home rehabilitation
- Treatment as usual (No Intervention): Patients will receive rehabilitation treatment after today's principles and routines.

INTERVENTIONS:
Other: Early supported discharge with day unit rehabilitation — Treatment by physiotherapist and occupational therapist up to 4 hours a day for up to 5 weeks in a day unit
  Arms: Day unit rehabilitation
Other: Early supported discharge with home rehabilitation — Treatment by physiotherapist and occupational therapist up to 4 hours a day for up to 5 weeks in the patient's home
  Arms: Home rehabilitation

SUMMARY:
The main purpose of this study is to evaluate the benefit of early supported discharge (ESD) in rehabilitation of stroke patients in two different outpatient modalities.

In a collaborating study, changes in physical function as well as the patients' own perception of physical function, pain and fatigue will be studied. In further collaborating studies, health economics and organizational issues will also be evaluated.

DETAILED DESCRIPTION:
Early supported discharge (ESD) seems to be at least as effective as hospital rehabilitation after stroke, and possibly better. In this study patients with recent stroke will be randomized to one of three different treatment arms:

* ESD with treatment at a day institution until 4 hrs. per day for up to 5 weeks
* ESD with treatment in the patients' home until 4 hrs. per day for up to 5 weeks
* Rehabilitation treatment "as usual", with a longer hospital stay, but without any specific treatment or follow-up after discharge

The patients in the two ESD arms will in addition be followed closely by a multidisciplinary coordinating team during the stay in hospital and the 5 week period of treatment after discharge, and they will be offered follow-ups at 3 and 6 months after inclusion into the study.

Patients in all 3 arms will be systematically examined with a set of measuring instruments as well as objective physical and function tests. This will be performed at inclusion and at 3, 6, 12 and 24 months after inclusion.

In the collaborating study by physiotherapist Bente Gjelsvik a comparison between changes in trunk control, balance, walking and ADL 3 months post stroke, as well as the patients' perceptions of physical function, pain and fatigue, will be the main focus. To assess function, functional change and possible differences between different interventions, there is a need for reliable and valid outcome measures. As a basis for the use of the outcome measure Trunk Impairment Scale (TIS) in this study, the TIS has been translated into Norwegian, Trunk Impairment Scale - Norwegian version (TIS-NV) and will be examined for measurement properties using data from the above study as well as data from patients with brain damage recruited from the Department of Physical Rehabilitation Medicine, Haukeland University Hospital. An examination of a possible connection between localisation and size of the stroke and trunk control will also be performed, as characteristics of the stroke may have therapeutic implications for the choice of intervention for the individual patient. The research questions for the planned doctoral thesis for Bente Gjelsvik are therefore as follows:

1. Is the TIS-NV reliable and valid in patients with brain damage?
2. Are changes in trunk control, balance, walking and daily activities, as well as pain and fatigue 3 months post stroke different in patients who have received interventions from different courses of rehabilitation in the study "Early supported discharge after stroke in Bergen"? To which degree do the patients perceive problems related to balance, physical activity, walking, pain and fatigue?
3. Is there a correlation between localization and size of the stroke as measured by magnetic tomography, and the patients' trunk control? Are initial localization and size of the stroke predictive for the patients' trunk control 3 months post stroke?

Another collaborating project is carried out by PhD candidate Hedda Døli (Language outcome after stroke: lesion location, prognosis and consequences).

The aim of her first study in the PhD project is to investigate the relationship between lesion location and aphasia severity one week post-stroke. Thereafter a follow-up study of the same patients 12 months post-stroke investigates the prognosis of aphasia and the variables that may influence recovery. In the third study the aim is to investigate the health-related quality of life and the occurrence of depression in patients with aphasia.

ELIGIBILITY:
Inclusion Criteria:

* Living in own home in the community of Bergen, Norway
* Inclusion within 1-7 days (24-168 hours) after debut of symptoms
* Inclusion within 6-120 hours after admission to Department of Neurology
* NIHSS score 2-26 at inclusion OR NIHSS score < 2 if Modified Rankin Scale is 2 or higher when being 0 before the stroke
* The patient must be awake and informed consent must be given by patient or relatives

Exclusion Criteria:

* Serious psychic illness
* Serious drug abuse
* Serious medical conditions that can influence the patients' cerebrovascular disease or rehabilitation
* Poor knowledge of the Norwegian language

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2008-12; Primary Completion 2012-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
MRS | 6 months
  Modified Rankin Scale

SECONDARY OUTCOMES:
NIHSS | 3, 6 and 12 months
  National Institutes of Health Stroke Scale
BI | 3, 6, 12 and 24 months
  Barthel ADL Index
AMPS | 3 and 6 months
  Assessment of Motor and Process Skills
TIS | 3 and 6 months
  Trunk Impairment Scale
SIS | 12 months
  Stroke Impact Scale
RSS | 12 months
  Relative Stress Scale
PGIC | 12 and 24 months
  Patients' Global Impression of Change
SF-36 | 12 and 24 months
  Short Form (36) Health Survey
MRS | 3, 12 and 24 months
  Modified Rankin Scale
PASS (Postural Assessment Scale for Stroke) | 3 and 6 months
5mTW (5 meter Timed Walk) | 3 and 6 months
TUG (Timed Up and Go) | 3 and 6 months
NRS (Numeric Rating Scale) | 3 and 6 months
Norwegian Basic Test for Aphasia | 3 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jan S. Skouen, PhD, Study Director — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Norway

REFERENCES:
- [Background] Hofstad H, Naess H, Moe-Nilssen R, Skouen JS. Early supported discharge after stroke in Bergen (ESD Stroke Bergen): a randomized controlled trial comparing rehabilitation in a day unit or in the patients' homes with conventional treatment. Int J Stroke. 2013 Oct;8(7):582-7. doi: 10.1111/j.1747-4949.2012.00825.x. Epub 2012 May 18. PMID 22594689
- [Result] Gjelsvik B, Breivik K, Verheyden G, Smedal T, Hofstad H, Strand LI. The Trunk Impairment Scale - modified to ordinal scales in the Norwegian version. Disabil Rehabil. 2012;34(16):1385-95. doi: 10.3109/09638288.2011.645113. Epub 2011 Dec 23. PMID 22191850
- [Derived] Hofstad H, Gjelsvik BE, Naess H, Eide GE, Skouen JS. Early supported discharge after stroke in Bergen (ESD Stroke Bergen): three and six months results of a randomised controlled trial comparing two early supported discharge schemes with treatment as usual. BMC Neurol. 2014 Dec 21;14:239. doi: 10.1186/s12883-014-0239-3. PMID 25528166
- [Derived] Gjelsvik BE, Hofstad H, Smedal T, Eide GE, Naess H, Skouen JS, Frisk B, Daltveit S, Strand LI. Balance and walking after three different models of stroke rehabilitation: early supported discharge in a day unit or at home, and traditional treatment (control). BMJ Open. 2014 May 14;4(5):e004358. doi: 10.1136/bmjopen-2013-004358. PMID 24833680